CLINICAL TRIAL: NCT03511326
Title: Subject Reported Outcomes on Satisfaction, Safety and Efficacy With Luxerm® in the Field-directed Treatment of Thin or Non-hyperkeratotic and Non-pigmented Actinic Keratosis of the Face or the Scalp
Brief Title: PRO With Luxerm® in the Field Treatment of Thin and Non-hyperkeratotic Non-pigmented AK
Acronym: SESAME 2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RD.03.SPR.114384
Record Dates: First submitted 2017-08-25; First posted 2018-04-27 (Actual); Results first posted 2020-12-10 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2018-09

CONDITIONS: Actinic Keratoses
Keywords: field-treatment
MeSH Terms: conditions — Keratosis, Actinic | interventions — methyl 5-aminolevulinate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Luxerm® (Experimental)
  Interventions: Drug: Methyl Aminolaevulinate 16% Cream

INTERVENTIONS:
Drug: Methyl Aminolaevulinate 16% Cream — Subject will received one session of methyl aminolevulinate Daylight Photodynamic therapy
  Other Names: 160mg/g of methyl aminolevulinate

SUMMARY:
Interventional open label prospective and multicentre study conducted in Germany in subjects with thin or non-hyperkeratotic and non-pigmented multiple AKs in one anatomical area on the face (e.g., forehead or cheek or chin), excluding nose eyelids, lips and mucosa or balding scalp, using Luxerm® DL-PDT treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age > 18 years old.
2. Subject with at least 5 clinically confirmed thin or non-hyperkeratotic and non-pigmented actinic keratoses in an anatomical area on the face (e.g., forehead or cheek or chin) excluding nose, eyelids, lips and mucosa, or balding scalp, at baseline visit.
3. Subject or caregiver capable of performing the skin preparation and Luxerm® treatment application as per the investigator instructions.
4. Female subject of childbearing potential must have a negative UPT at baseline (UPT should have a sensitivity of 25 IU/L or less) and agree to be strictly abstinent or use a highly effective method of birth control during the study (i.e. progestogen-only oral hormonal contraception; male or female condom; cap, diaphragm or sponge with spermicide; bilateral tubal ligation; combined (estrogen and progestogen-containing) oral hormonal contraception, or injectable or implants hormonal contraception (at a stable dose for at least 1 month prior to baseline); intra-uterine devices inserted at least 1 month prior to baseline; vasectomized partner for at least 3 months prior to baseline).
5. Female subject of non-childbearing potential, e.g.: post-menopausal (absence of menstrual bleeding for 1 year without any other medical reason), hysterectomy or bilateral ovariectomy.
6. Subject has read and signed the approved informed consent form (ICF) prior to any participation in the study.
7. Subject has read and signed a Photograph Release Consent Form if he/she is willing to be photographed.
8. Subject (or caregiver) willing and able to comply with all of the time commitments and procedural requirements of the clinical trial protocol.

Exclusion Criteria:

1. Subject with a clinical diagnosis of a skin disease other than AK (including non-melanoma skin cancer) on the target anatomical area.
2. Subject with severe AK (thick, hyperkeratotic AK) per anatomical area (face or scalp).
3. Subject with clinical diagnosis of other skin disease on the target anatomical area.
4. Subject with pigmented AK on the target anatomical area.
5. Subject with melanoma at any location.
6. Immunocompromised subject or requiring immunosuppressive therapies.
7. Subject with porphyria; photosensitivity- related disorders, active infectious disease.
8. Subject with known or suspected hypersensitivity to the active substance or to any excipients of Luxerm® (see Summary of Product Characteristics).
9. Female subject who is pregnant, nursing or planning a pregnancy during the study.
10. Subject who has used any of the following topical preparations on the area to be treated: keratolytics including urea (greater than 5%), alpha hydroxyacids [e.g. glycolic acid, lactic acid, etc. greater than 5%], salicylic acid (greater than 2%) within 2 days of initiation of treatment.
11. Subject with a wash-out period from baseline for topical or systemic treatment or medical/surgical procedure in the anatomical area (for AKs) less than the following:

    * Retinoids, including tazarotene, adapalene, tretinoin, retinol ==> 4 weeks
    * Cryotherapy, diclofenac, corticosteroids or other treatments for AK==> 8 weeks
    * Microdermabrasion, laser ablative treatments or chemical peels ==>8 weeks
    * 5-FU, imiquimod ==>24 weeks
    * Surgical: excision and reconstructive surgery, chemosurgery, ==>12 weeks
    * Any Photodynamic Therapy, ingenol mebutate (Pep-005), Radiotherapy and UV radiation therapy==>12 weeks
    * Investigational therapies for Actinic Keratoses==>12 weeks
    * Immunosuppressive drugs (such as glucocorticoids, cytostatic, antibodies, drugs acting on interferon, opioids, TNF binding proteins, Mycophenolate, small biologics agents)==>12 weeks
12. Subject who is currently participating to/ or who has participated in another investigational treatment or device research study within 4 weeks of baseline visit.
13. Subject may be unreliable for the study including subjects who engage in excessive alcohol intake or drug abuse, or subjects who are unable to return for scheduled follow-up visits.
14. Subject who is unable to communicate or cooperate with the investigator due to language problems, poor mental development, or impaired cerebral function.
15. Subject who is unwilling to refrain from use of prohibited medication during the clinical trial (see section 4.3.5).
16. Subject who is vulnerable (such as deprived of freedom) as defined in Section 1.61 of the International Conference on Harmonisation (ICH) Guideline for Good Clinical Practice (GCP).
17. Subject with clinically significant abnormal laboratory finding (if any available report) at the baseline visit or medical/surgical condition (other than for actinic keratoses), which might, in the Investigator's opinion, interfere with study evaluations or pose a risk to subject safety during the study.
18. The subject is a study site staff member (investigator, study nurse, etc.) or a relative of one.
19. Subjects with any condition that may be associated with a risk of poor protocol compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-06-07 (Actual); Primary Completion 2017-11-28 (Actual); Study Completion 2017-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajeev CHAVDA, MD, Study Director — Galderma R&D
Locations (1):
- University Hospital Regensburg, Regensburg, Germany

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Luxerm®
Started | 50
Completed | 49
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Luxerm®
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.4 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 50
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Germany | 50
Skin phototype [Count of Participants; unit: Participants] — Fitzpatrick skin phototype is a system used to describe a person's skin type. It ranges from skin phototype I to III. Where, skin phototype I = pale white skin, always burns easily, never tans; skin phototype II = fair skin, always burns easily, tans minimally and with difficulty; skin phototype III = darker white skin, burns minimally, tans gradually and uniformly.
  Participants
    Phototype I | 7
    Phototype II | 35
    Phototype III | 8
Duration of Actinic Keratosis [Mean (Standard Deviation); unit: years] | 7.77 (6.78)

OUTCOME MEASURES:

1. Primary Outcome: Overall Subject Satisfaction the Day of Treatment After Daylight Session
Description: Percentage of subjects satisfied and very satisfied globally with Luxerm Daylight procedure, the day of treatment after daylight session
Time Frame: the day of treatment after daylight session
Population: Intent to Treat (ITT) population included all enrolled participants (i.e. treatment dispensed).
Measure: Count of Participants; unit: Participants
Arm/Group | Luxerm®
Number analyzed (Participants) | 50
Participants | 47

2. Primary Outcome: Overall Subject Satisfaction at Week 12 Post-treatment
Description: Percentage of subjects satisfied or very satisfied (overall) with Luxerm DL procedure
Time Frame: Week 12
Population: ITT population included all enrolled participants (i.e. treatment dispensed). Here, the "N" number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Luxerm®
Number analyzed (Participants) | 48
Participants | 41

ADVERSE EVENTS:
Time Frame: From signing of Informed Consent Form (ICF) to end of study (Week 12)
Arm/Group | Luxerm®
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 28/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Luxerm® (N=50)
Procedural pain (Injury, poisoning and procedural complications) | 15 (15)
Erythema (Skin and subcutaneous tissue disorders) | 19 (20)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 8 (8)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin tightness (Skin and subcutaneous tissue disorders) | 1 (1)
Skin warm (Skin and subcutaneous tissue disorders) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-22): https://cdn.clinicaltrials.gov/large-docs/26/NCT03511326/Prot_SAP_000.pdf